CLINICAL TRIAL: NCT05770115
Title: A Randomized Clinical Study Based on Comparison Between Closure of Uterine Incision With Vicryl 2/0 Versus Vicryl 1 in Development of Uterine Niche.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassiony Dabian, lecturer of obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MS-467-2020
Record Dates: First submitted 2023-01-29; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Cesarean Section; Dehiscence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): vicryl 2/0
  Interventions: Procedure: Vicryl 2/0
- Group B (Active Comparator): vicryl 1
  Interventions: Procedure: Vicryl 1

INTERVENTIONS:
Procedure: Vicryl 1 — Double layer closure with split thickness with vicryl 1, in continuous, non-locked, 1 cm apart sutures.
  Arms: Group B
Procedure: Vicryl 2/0 — Double layer closure with split thickness with vicryl 2/0, in continuous, non-locked, 1 cm apart sutures.
  Arms: Group A

SUMMARY:
The first group patients underwent double layer closure with split thickness with vicryl 2/0, in continuous, non- locked, 1 cm apart sutures, study group, and the second group, women underwent double layer closure with split thickness with vicryl 1, in continuous, non- locked, 1 cm apart sutures, control group. Then, all women in the study were followed up for development of niche within 1 to 6 weeks. The assessment after one week postpartum was with using trans-abdominal Ultrasound, then after two to six weeks postpartum with transvaginal Ultrasound

DETAILED DESCRIPTION:
Caesarean section rates have increased worldwide over the past decades from 6.7 to 19.1%, with a current European CS rate of 25% of all births. CS is considered to be a safe procedure that can be life saving for both mother and child but the increasing trend draws more attention to adverse outcomes related to CSs. A relatively new long-term sequela is the niche in the uterine caesarean scar. A niche is defined as "an indentation at the site of the uterine caesarean scar with a depth of at least 2 mm on ultrasound" and is present in 56-84% of women after one or more CSs .

It is realized that almost all of the increase in cesarean section rate is due to the increase in repeat operations, and primary cesarean deliveries for dystocia and fetal distress. These can be attributed to obstetric factors as increased primary cesarean delivery rate, failed induction. Maternal factors as Increased proportion of women > age 35, increased nulliparous women, increased elective primary cesarean deliveries and factors relating to the physician as Malpractice litigation concerns .

The hypotheses can be divided into surgery-related factors and patient related factors. In their paper they focused on surgery-related factors since these could be easily modified and studied in future RCTs .

These surgical-related factors include low (cervical) location of the uterine incision during a CS, Incomplete closure of the uterine wall, due to single-layer, endometrial saving closure technique or use of locking sutures and Surgical activities that may induce adhesion formation (i.e., non-closure of peritoneum, inadequate hemostasis, applied sutures, use of adhesion barriers).

Without questions, the uterine niche presents a pathology that requires evaluation and intervention to mitigate its prevalence. The aim of this study is to compare between closures of uterine incision with Vicryl 2/0 versus Vicryl 1 in developing a uterine niche.

ELIGIBILITY:
Inclusion Criteria:

* Singleton term pregnancy.
* Parity less than 5.
* Women who undergo 1st cesarean section whether in labor or not.

Exclusion Criteria:

* Women with a previous CS.
* Previous major uterine surgery (e.g. laparoscopic or laparotomic fibroid resection, septum resection).
* Women with known causes of menstrual disorders (e.g. cervical dysplasia, communicating hydro-salpinx, uterine anomaly or endocrine disorders disturbing ovulation).
* Abnormally invasive placenta during the current pregnancy.
* Multiple gestation, polyhydramnios.
* Maternal Diabetes, anemia and connective tissue disorders.
* Women with Body mass index > 35.
* Women with valval varicosities.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 264 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
prevalence of uterine niche | 6 weeks
  using transvaginal ultrasound for detection of development of CS scar niche

SECONDARY OUTCOMES:
operative time | 1 hour
  operative time in minutes is measured from the time of skin incision to time of skin closure
size of cs niche | 6 weeks
  size of cs niche is measured in millimeters using transvaginal ultrasound.
operative blood loss | 2 hours
  operative blood loss in milliliteres as indicated by the wieghing the towels before and after CS.
postoperative haemoglobin | 24 hours
  measured in mg/dl as full blood count is done 24 hours postoperative.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy outpatient infertility clinic, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bij de Vaate AJ, van der Voet LF, Naji O, Witmer M, Veersema S, Brolmann HA, Bourne T, Huirne JA. Prevalence, potential risk factors for development and symptoms related to the presence of uterine niches following Cesarean section: systematic review. Ultrasound Obstet Gynecol. 2014 Apr;43(4):372-82. doi: 10.1002/uog.13199. PMID 23996650
- [Background] Byrne M, Aly A. The Surgical Suture. Aesthet Surg J. 2019 Mar 14;39(Suppl_2):S67-S72. doi: 10.1093/asj/sjz036. PMID 30869751
- [Background] 70. Monika & Gupta, Monika & Goraya, s.P.s & Kaur, Tanjeet & Matreja, Prithpal. (2017). Single Layer Versus Double Layer Closure of Uterus during Caesarean Section - A Prospective Study in Index and Subsequent Pregnancy. International Archives of BioMedical and Clinical Research. 1. 10.21276/iabcr.2017.3.1.14.